CLINICAL TRIAL: NCT04799405
Title: Supervised Home-based Transcranial Direct Current Stimulation (tDCS) for Major Depressive Disorder
Brief Title: Home-based tDCS in Major Depressive Disorder
Acronym: MoodStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Senior Scientist-Professor of Neurology, Hebrew SeniorLife
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00044198
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
Keywords: non-invasive brain stimulation (NIBS); transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- tDCS MDD (Experimental): A group of 5 participants with major depressive disorder (MDD).
  tDCS, as a relatively simple and portable technology, is particularly well suited for remotely-supervised, home-based treatment, which would facilitate longer periods of treatment as well as offer a suitable therapeutic option at the present time as the investigators aim to deal with the COVID-19 pandemic.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Daily sessions (28 daily sessions): The device will be used to apply 30 minutes of tDCS to the participant with MDD's scalp in each of 28 daily sessions.
  Thereafter, participants with MDD will undergo a taper phase of an additional 9 sessions of tDCS applied in progressively decreasing frequency until day #60 of the study as follows:
  1. First taper phase: three 30 minutes tDCS sessions applied every other day;
  2. Second taper phase: three 30 minutes tDCS sessions applied one every third day;
  3. Third and final taper phase: three final 30 minutes tDCS sessions applied one every fourth day.
  Other Names: Transcranial direct current stimulation (tDCS)

SUMMARY:
The investigators propose a study of telehealth supervised, caregiver-delivered, home-based transcranial direct current stimulation (tDCS) for antidepressant treatment of patients with an acute depressive episode.

DETAILED DESCRIPTION:
This is an open-label pilot feasibility telemedicine study. This pilot will involve a total of 37 stimulations sessions / at home visits (30- minute sessions of multichannel excitatory tDCS targeting the left DPFC) and the maintenance of a daily treatment diary to be completed by the subjects immediately after enrollment and 12 weeks following the last study visit.

ELIGIBILITY:
Patients meeting one of the following criteria may be eligible to participate in this study.

1. Patients with medication-resistant MDD who have undergone rTMS or ECT and responded to it but whose benefit has lapsed, and they need repeat a rTMS or ECT course that they cannot access
2. Patients with medication-resistant MDD who have undergone rTMS or ECT and responded to it but whose benefit has lapsed, and they need repeat a rTMS or ECT course that they cannot access
3. Patients with medication-resistant MDD who are undergoing rTMS or ECT and responding, but cannot continue to get the rTMS or ECT course due to COVID-19 pandemic-related regulations or other access concerns
4. Patients with medication-resistant MDD who are referred to rTMS or ECT and are found well qualified but cannot access rTMS or ECT due to COVID-19 pandemic-related regulations or other access concerns.

The benefits of this project address a present need due to the COVID-19 pandemic, but also go beyond the present situation and address a larger, pre-existing need. Across all these potential groups of participants, prospective participants will:

* need to have a primary psychiatrist who agrees to their participation in the study and is willing to continue to follow the patient and work collaboratively with the study team
* need to be assessed by their primary psychiatrist to be stable enough to be able to remain at home and participate in the present study without undue risk to their safety
* need to be living with an adult willing and capable to provide oversight and learn to deliver the home-based tDCS
* have the capability to connect with the study team for daily supervision of the intervention sessions and close safety monitoring, and be willing to commit to doing so

Inclusion Criteria:

Individuals with MDD

Participants will be men and women who:

* Are aged 50 or older
* Able to read, write, and communicate in English
* Have a caregiver who is willing and able to provide the home tDCS sessions.
* Participants must be under the care of a treating psychiatrist who approves of the study participation and believes that TMS or ECT is indicated for his/her patient but that

  * it would not endanger the patient to participate in the present study rather than pursue such alternative, or
  * the patient could not gain access to TMS or ECT due to COVID-19 (The depression phase of bi-polar disorder is not a reason for exclusion if the treating psychiatrist believes TMS or ECT would be indicated).

Participants with MDD must fit into one of the following 3 groups (medication-resistant MDD defined as 1) participant's condition has not responded to prescribed antidepressant medication; 2) participant is medication intolerant, or 3) some other underlying reason):

* Patients with medication-resistant Major depressive disorder (MDD) who have undergone repetitive transcranial magnetic stimulation (rTMS) or electroconvulsive therapy (ECT) and responded to it but whose benefit has lapsed and they need repeat rTMS or ECT course that they cannot access;
* Patients with medication-resistant MDD who are undergoing rTMS or ECT and responding, but cannot continue to get the rTMS or ECT course due to COVID-19 pandemic-related regulations or other access concerns
* Patients with medication-resistant MDD who are referred to rTMS or ECT and are found well qualified but cannot access rTMS or ECT due to COVID-19 pandemic-related regulations or other access concerns.

Further, participants must:

* Meet criteria for a diagnosis of MDD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) (American Psychiatric Association, 2000), as determined via an tele-health interview with a study psychiatrist, and confirmed with the Mini International Neuropsychiatric Interview (MINI; Version 5.0.0) (Sheehan et al., 1998) and the prospective participant's primary psychiatrist.
* Currently experiencing a major depressive episode of at least four weeks' duration as part of a unipolar or bipolar depression. Score will need to be at least 20 on the MADRS.

Further, participants must have a willing and eligible caregiver-administrators who is:

* At least 21 years of age
* Able to read, write, and communicate in English
* Self-reported computer proficiency and willingness to learn how to use tDCS as defined by "yes" answers to the questions "Do you feel comfortable using a computer?" and "are you willing to learn
* How to administer tDCS?" Stated availability throughout the study period to administer tDCS sessions to the participant with MDD.

Exclusion Criteria:

* Exclusion criteria for participants with MDD will be:

  * Any DSM-psychotic disorder
  * Drug or alcohol abuse or dependence in the preceding three months;
  * Concurrent benzodiazepine medication;
  * High suicide risk (Utilizing the Beck Depression Inventory and the Hamilton Depression Scale, suicide risk will be assessed at baseline by the study psychiatrist) ;
  * History of clinically defined neurological disorder or insult; Metal in the cranium or skull defects;
  * Skin lesions on the scalp at the proposed electrode sites;
  * Pregnancy.
  * Medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagus nerve stimulator).
  * Previous skull surgery with resultant skull defects
  * Inability to understand study procedures following review of the Informed Consent form.

Understanding will be assessed by asking the participant with MDD to answer the following three questions:

1. What is the purpose of this study?
2. What are the risks of study involvement?
3. If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form. Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Exclusion criteria for Participant caregiver-administrators:

* Poor eyesight,
* Severe arthritis in the hands, pain, deformity or other condition that interferes with successful administration of tDCS.
* Inability to understand study procedures following review of the Informed Consent form.

Understanding will be assessed by asking the participant caregiver-administrator to answer the following three questions:

1. What is the purpose of this study?
2. What are the risks of study involvement?
3. If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form (see attached). Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, Dr., Principal Investigator — Hinda and Arthur Marcus Institute for Aging Research
Locations (1):
- Hinda and Arthur Marcus Institute for Aging Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alonzo A, Fong J, Ball N, Martin D, Chand N, Loo C. Pilot trial of home-administered transcranial direct current stimulation for the treatment of depression. J Affect Disord. 2019 Jun 1;252:475-483. doi: 10.1016/j.jad.2019.04.041. Epub 2019 Apr 10. PMID 31005790
- [Result] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Result] Brunoni AR, Moffa AH, Fregni F, Palm U, Padberg F, Blumberger DM, Daskalakis ZJ, Bennabi D, Haffen E, Alonzo A, Loo CK. Transcranial direct current stimulation for acute major depressive episodes: meta-analysis of individual patient data. Br J Psychiatry. 2016 Jun;208(6):522-31. doi: 10.1192/bjp.bp.115.164715. Epub 2016 Apr 7. PMID 27056623
- [Derived] Cappon D, den Boer T, Jordan C, Yu W, Lo A, LaGanke N, Biagi MC, Skorupinski P, Ruffini G, Morales O, Metzger E, Manor B, Pascual-Leone A. Safety and Feasibility of Tele-Supervised Home-Based Transcranial Direct Current Stimulation for Major Depressive Disorder. Front Aging Neurosci. 2022 Feb 2;13:765370. doi: 10.3389/fnagi.2021.765370. eCollection 2021. PMID 35185515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events occurred between participant enrollment and start of the intervention.
Groups:
- tDCS MDD: A group of participants with major depressive disorder (MDD).
  tDCS, as a relatively simple and portable technology, is particularly well suited for remotely-supervised, home-based treatment, which would facilitate longer periods of treatment as well as offer a suitable therapeutic option at the present time as the investigators aim to deal with the COVID-19 pandemic.
  tDCS: Daily sessions (28 daily sessions): The device will be used to apply 30 minutes of tDCS to the participant with MDD's scalp in each of 28 daily sessions.
  Thereafter, participants with MDD will undergo a taper phase of an additional 9 sessions of tDCS applied in progressively decreasing frequency until day #60 of the study as follows:
  1. First taper phase: three 30 minutes tDCS sessions applied every other day;
  2. Second taper phase: three 30 minutes tDCS sessions applied one every third day;
  3. Third and final taper phase: three final 30 minutes tDCS sessions applied one every fourth day.
Period: Phase 1 - Acute Stimulation, Daily tDCS
Arm/Group | tDCS MDD
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Phase 2 - Tapered Stimulation Schedule
Arm/Group | tDCS MDD
Started | 3
Completed | 3
Not Completed | 0
Period: Phase 3 - Follow up Phase
Arm/Group | tDCS MDD
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- tDCS MDD: A group of 5 participants with major depressive disorder (MDD).
  tDCS, as a relatively simple and portable technology, is particularly well suited for remotely-supervised, home-based treatment, which would facilitate longer periods of treatment as well as offer a suitable therapeutic option at the present time as the investigators aim to deal with the COVID-19 pandemic.
  tDCS: Daily sessions (28 daily sessions): The device will be used to apply 30 minutes of tDCS to the participant with MDD's scalp in each of 28 daily sessions.
  Thereafter, participants with MDD will undergo a taper phase of an additional 9 sessions of tDCS applied in progressively decreasing frequency until day #60 of the study as follows:
  1. First taper phase: three 30 minutes tDCS sessions applied every other day;
  2. Second taper phase: three 30 minutes tDCS sessions applied one every third day;
  3. Third and final taper phase: three final 30 minutes tDCS sessions applied one every fourth day.
Arm/Group | tDCS MDD
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Full Range); unit: units on a scale] — The MADRS is a clinician-rated scale which consists of 10 items; each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points, with higher scores indicative of greater depressive symptomology (Montgomery & Åsberg, 1979). The primary outcome was the change in the MADRS score from baseline to the 1-month follow-up (12 week span). Remission was defined as MADRS score ≤ 10.
  units on a scale | 35 [27 to 44]
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) [Mean (Full Range); unit: units on a scale] — The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item questionnaire that captures life satisfaction over the past week across several domains. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). The Total Score is reported as percentage maximum possible % Max = Raw-minimum score/maximum score-minimum score.
  units on a scale | 33.2 [30 to 36]
Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report)(QIDS-SR16) [Mean (Full Range); unit: units on a scale] — The Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report)(QIDS-SR16) is a self-report measure of depressed symptomology. Questions in the QIDS - SR-16 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance, Sad mood,The total score ranges from 0 to 27.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
  units on a scale | 17.6 [12 to 26]
Beck Depression Inventory (BDI) [Mean (Full Range); unit: units on a scale] — The Beck Depression Inventory (BDI) is 21-item multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. For each item, a value of 0 to 3 is assigned and then the total score is summed. The standard cut-offs are as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
  units on a scale | 24.8 [17 to 36]
Hamilton Depression Rating Scale (HDRS) [Mean (Full Range); unit: units on a scale] — Hamilton Depression Rating Scale (HDRS) is comprised of 21 items for inquiry, and only the first 17 are used in scoring. Each question examines a different symptom or aspect of depression, including: mood, guilt, suicidal ideation, insomnia, agitation, and somatic symptoms. Items are scaled either from 0 - 2 or 0 - 4, and each item is summed for a total score. Benchmarks suggested at: 0-7 normal; 8 - 13 mild depression; 14-18 moderate depression; 19-22 severe depression ; >=23 very severe depression.
  This scale was administered at baseline and 12 weeks later at the 1-month follow-up visit.
  units on a scale | 19.8 [14 to 24]
Montreal Cognitive Assessment (MoCA) [Mean (Full Range); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains. The total possible score is 30 points; a score of 26 or above is considered normal. Severity of impairment can be determined with the following scores: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment, and less than 10= severe cognitive impairment. The maximum total score is 30 and the minimum total score is 0 points.
  This assessment was administered at baseline and at 1 month post-intervention (12 week span).
  units on a scale | 27.8 [22 to 30]
Digit Span Forward [Mean (Full Range); unit: Count of numbers correctly recalled] — A digit-span forward task measures working memory storage capacity of numbers. Participants are auditorily presented with a chain of numerical digits and are instructed to recall the sequence of numbers verbally in the order that it was presented to the participant. The number of digits on the first trial is three. The length of the sequence increases with each correct trial completion. The more numbers recalled the better a participants has done.
  Count of numbers correctly recalled | 7.6 [6 to 9]
Digit Span Backward [Mean (Full Range); unit: Count of numbers correctly recalled] — A digit-span task backwards measures working memory storage capacity of numbers. Participants are auditorily presented with a chain of numerical digits and are instructed to recall the sequence of numbers verbally in backwards order. The number of digits on the first trial is two. The length of the sequence increases with each correct trial completion. The more numbers recalled the better a participants has done.
  Count of numbers correctly recalled | 6 [4 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item clinical rating scale to measure the severity of depressive symptoms based on a clinical interview with a participant/patient. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60, and includes questions related to: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Cut off points are: 0 to 6 - normal, symptom absent, 7 to 19 - mild depression, 20 to 34 - moderate depression, >34 - severe depression. Clinical remission is considered as a MADRS score ≤ 10.
  The primary outcome will be total MADRS score from baseline to one-month follow-up (pre and post-intervention; 12 weeks).
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 16 [6 to 25]

2. Primary Outcome: Number of Treatment-Emergent Adverse Events [Safety and Tolerability] and Missed Sessions
Description: Feasibility and tolerability/safety will be evaluated using home-based data as recorded in the Neuroelectrics portal: number of missed sessions and number of adverse events reported on adverse event questionnaire
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Number; unit: number of sessions/events
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
number of sessions/events
  Number of missed sessions | 1
  Number of treatment-emergent adverse events | 0

3. Secondary Outcome: The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item questionnaire that captures life satisfaction over the past week across several domains. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). The Total Score is reported as percentage maximum possible % Max = Raw-minimum score/maximum score-minimum score. (Raw score minus the minimum possible raw score divided by the maximum possible raw score minus the minimum possible raw score).
  This measure was administered at baseline and at 1 month follow-up, which were separated by 12 weeks.
Time Frame: 12 weeks
Population: A group of participants with Major Depressive Disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 44.6667 [42 to 48]

4. Secondary Outcome: The Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report)(QIDS-SR16)
Description: The Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report)(QIDS-SR16) is a self-report measure of depressed symptomology. Questions in the QIDS - SR-16 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia) (Q 1 - 4), Sad mood (Q 5), Decrease/increase in appetite/weight (Q 6 - 9), Concentration (Q 10), Self-criticism (Q 11), Suicidal ideation (Q 12), Interest (Q 13), Energy/fatigue (Q 14), Psychomotor agitation/retardation (Q 15 - 16). Severity of depression can be judged based on the total score, which ranges from 0 to 27.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
  This measure was administered at baseline and at 1 month follow-up, which were separated by 12 weeks.
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 5.3333 [0 to 10]

5. Secondary Outcome: Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory (BDI) is 21-item multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. For each item, a value of 0 to 3 is assigned and then the total score is summed. The standard cut-offs are as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
  This scale was given at baseline and 12 weeks later at the 1-month follow-up visit.
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 10.3333 [2 to 18]

6. Secondary Outcome: Hamilton Depression Rating Scale
Description: Hamilton Depression Rating Scale (HDRS) is comprised of 21 items for inquiry, and only the first 17 are used in scoring. Each question examines a different symptom or aspect of depression, including: mood, guilt, suicidal ideation, insomnia, agitation, and somatic symptoms. Items are scaled either from 0 - 2 or 0 - 4, and each item is summed for a total score. Benchmarks suggested at: 0-7 normal; 8 - 13 mild depression; 14-18 moderate depression; 19-22 severe depression ; >=23 very severe depression.
  This scale was administered at baseline and 12 weeks later at the 1-month follow-up visit.
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 7.3333 [1 to 14]

7. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) is designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains. The total possible score is 30 points; a score of 26 or above is considered normal. Severity of impairment can be determined with the following scores: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment, and less than 10= severe cognitive impairment. The maximum total score is 30 and the minimum total score is 0 points.
  This assessment was administered at baseline and at 1 month post-intervention (12 week span).
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
units on a scale | 28.6667 [28 to 30]

8. Secondary Outcome: Digit Span Forward
Description: A digit-span forward task measures working memory storage capacity of numbers. Participants are auditorily presented with a chain of numerical digits and are instructed to recall the sequence of numbers verbally in the order that it was presented to the participant. The number of digits on the first trial is three. The length of the sequence increases with each correct trial completion. The more numbers recalled the better a participants has done.
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: Count of numbers correctly recalled
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
Count of numbers correctly recalled | 8 [7 to 9]

9. Secondary Outcome: Digit Span Backward
Description: A digit-span task backwards measures working memory storage capacity of numbers. Participants are auditorily presented with a chain of numerical digits and are instructed to recall the sequence of numbers verbally in backwards order. The number of digits on the first trial is two. The length of the sequence increases with each correct trial completion. The more numbers recalled the better a participants has done.
Time Frame: 12 weeks
Population: A group of participants with major depressive disorder (MDD).
Measure: Mean (Full Range); unit: Count of numbers correctly recalled
Arm/Group | tDCS MDD
Number analyzed (Participants) | 3
Count of numbers correctly recalled | 6 [4 to 8]

ADVERSE EVENTS:
Time Frame: 6 months
Description: It does not differ.
Arm/Group | tDCS MDD
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT04799405/Prot_SAP_000.pdf